CLINICAL TRIAL: NCT07219459
Title: A Phase 2b, Randomized, Blinded Trial Investigating the Efficacy and Safety of Visugromab in Combination With Nivolumab and a Tyrosine Kinase Inhibitor Compared to Double Placebo and a Tyrosine Kinase Inhibitor in Participants With Unresectable or Metastatic Hepatocellular Carcinoma and Compensated Liver Function (Child-Pugh A) After Failure of First-Line Treatment That Included an Anti PD-(L)1 Compound (GDFATHER HCC-01)
Brief Title: Visugromab, Nivolumab and a Tyrosine Kinase Inhibitor (TKI) Compared to Double Placebo and a TKI in Unresectable or Metastatic Hepatocellular Carcinoma Post Anti-PD-(L)1 Failure
Acronym: GDFATHERHCC01
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CatalYm GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTL-002-005; 2025-520675-86-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-20; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Unresectable or Metastatic Hepatocellular Carcinoma; Failure of First-Line Treatment That Included an Anti PD-(L)1 Compound; Child-Pugh A Hepatocellular Carcinoma
Keywords: CTL-002; Visugromab; GDF-15
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab; Tyrosine Kinase Inhibitors; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Throughout the randomized, blinded, placebo-controlled part (Part 2) of the trial, the participants, Investigators, and trial assigned site staff (except for the pharmacists), the clinical CRO (except for the unblinded clinical monitoring team), and imaging vendor will remain blinded to the information which participant is receiving which IMP. The biostatistics provider, central laboratory vendor, safety vendor and Sponsor also remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Visugromab (IV) + Nivolumab intravenous (IV) + TKI (PO)
  Interventions: Biological: Visugromab RDE (recommended dose for expansion); Biological: Nivolumab; Drug: Tyrosine kinase inhibitor (TKI)
- Arm B (Active Comparator): TKI (PO) + saline (double-placebo) intravenous (IV)
  Interventions: Drug: Tyrosine kinase inhibitor (TKI); Other: Placebo Saline Infusion

INTERVENTIONS:
Biological: Visugromab RDE (recommended dose for expansion) — Participants receive visugromab (RDE) intravenous (IV) on Day 1 of every 21-day cycle (every 3 weeks, or Q3W) for up to 35 treatments
  Other Names: CTL-002
  Arms: Arm A
Biological: Nivolumab — Participants receive Nivolumab 360mg intravenous (IV) on Day 1 of every 21-day cycle (every 3 weeks, or Q3W) for up to 35 treatments after visugromab infusion
  Other Names: OPDIVO®
  Arms: Arm A
Drug: Tyrosine kinase inhibitor (TKI) — Participants receive the TKI (PO)
Other: Placebo Saline Infusion — Saline (0.9%NaCl) intravenous (2x IV) on Day 1 of every 21-day cycle every 3 weeks (Q3W) for up to 35 treatments
  Other Names: 0.9% NaCl
  Arms: Arm B

SUMMARY:
This is a Phase 2b, randomized, blinded clinical trial investigating the efficacy and safety of visugromab in combination with nivolumab and a TKI compared to double placebo and a TKI in participants with unresectable or metastatic HCC and compensated liver function (Child-Pugh A) after failure of 1L treatment that included an anti-PD-(L)1 compound. The trial consists of 2 Parts: a non-randomized Safety-run-in part (Part 1) and the subsequent randomized part (Part 2) with 2 treatment arms (A and B). Randomization of participants into Treatment Arm A and B will continue until 40 efficacy-evaluable participants are enrolled into each Treatment Arm.

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically confirmed diagnosis of unresectable or metastatic HCC, not amenable to a curative treatment approach.
* Measurable disease as per RECIST v1.1 as determined by the Investigator based upon local radiologist assessment.
* Must have failed one line of prior systemic treatment for unresectable or metastatic HCC containing an approved anti PD (L)-1 checkpoint inhibitor (CPI) with a minimum treatment duration of 12 weeks exposure for the CPI with no documented progression in this period.
* Age ≥ 18 years on the day of signing the informed consent.
* Life expectancy of at least 3 months as assessed by the Investigator.
* ECOG performance status ≤1.
* Child-Pugh score of A6 or better.

Main Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC or mixed cholangiocarcinoma.
* More than 1 line of prior systemic treatment for unresectable or metastatic HCC.
* Received or completed any palliative radiotherapy for symptoms within 28 days of the first dose of IMP.
* Expected to require any other form of antineoplastic therapy during the trial.
* Clinically active inflammatory bowel disease, active diverticulitis, intra-abdominal abscess, and/or gastrointestinal obstruction.
* Known history of other prior malignancy unless participant has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.
* Known or detected clinically active central nervous system (CNS) involvement by HCC or other tumors.
* Have one of the following cardiovascular risk factors: myocardial infarction, peri/myocarditis, or history of ischemic stroke in the past 3 months before planned treatment start, uncontrolled heart failure, uncontrolled ventricular arrhythmia, QT interval corrected for heart rate using Fridericia's formula interval ≥ 470 ms regardless of sex.
* An active autoimmune disease that has required systemic treatment in past 3 months before planned treatment start.
* Comedication with metformin or metformin-containing antidiabetics in participants with type II diabetes.
* Chronic systemic corticosteroid treatment for other reasons.
* Prior liver or other organ transplantation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 36 months
  Investigator assessed Progression-free survival (PFS) time from randomization (during Safety Run-In: initiation of treatment) to first documented disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
Independently assessed PFS by Blinded Independent Central Review (BICR) | up to 36 months
CR (Complete Response) rate | up to 36 months
PR (Partial Response) rate | up to 36 months
ORR (Overall Response) rate | up to 36 months
  Overall response rate, defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) per RECIST v1.1 as assessed by the Investigator
TTR (Time-to-response) rate | up to 36 months
PFS (Progression-free survival) rate | up to 36 months
Participant weight course over time | up to 39 months
Adverse Events | up to 60 months
  Incidence, type and severity of adverse events, treatment emergent adverse events, treatment-related adverse events and serious adverse events
European Organization for Research and Treatment of Cancer quality-of-life questionnaire for cancer (EORTC QLQ-C30) | up to 39 months
  Assess participants' subjective wellbeing
Overall survival (OS) | up to 60 months

OTHER OUTCOMES:
Maximum concentration (Cmax) of visugromab | At designated time points (up to 36 months)
  Cmax is the maximum observed serum concentration of visugromab
Minimum concentration (Cmin) of visugromab | At designated time points (up to 36 months)
  Cmin is the minimum observed serum concentration of visugromab
Functional Assessment of the Anorexia and Cachexia Therapy questionnaire (FAACT-A/CS) | up to 39 months
  FAACT-ACS consists of 12 items assessing anorexia/cachexia-related symptoms. Each item is scored individually from 0 ("Not at all") to 4 ("Very much"), with some requiring reverse scoring as in the FAACT Scoring Guideline. The FAACT-ACS subscale score is calculated by summing item scores (reversals performed as applicable); multiplied by the total number of items and divided by the number of items answered. The total score ranges from 0-48, with higher scores indicating better anorexia/cachexia-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No